CLINICAL TRIAL: NCT06729112
Title: Pan-immune-inflammation Value (PIN) in Behçet's Disease and Its Correlation With Disease Activity
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Farrag Ahmed Mohamed, Lecturer of Rheumatology and Rehabilitation, Assiut University
Other Study IDs: SFA122024
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Behçet's disease: Adult Behçet's disease patients who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease.
  and Accept to participate in the current study.
  Interventions: Diagnostic Test: pan immune inflammation value
- control group: healthy matched controls
  Interventions: Diagnostic Test: pan immune inflammation value

INTERVENTIONS:
Diagnostic Test: pan immune inflammation value — Using the ratio of neutrophil, monocyte, and platelet counts to lymphocyte count, NLR, MLR, and PLR were calculated. The pan immune inflammation value (PIV) was calculated by multiplying the neutrophil count by the platelet count and the monocyte count, and then dividing the result by the lymphocyte count.

SUMMARY:
Behçet's disease (BD) is a systemic vasculitis affecting both small and large blood vessels in the venous and arterial systems. It is a multiorgan disease with various manifestations, including mucocutaneous, articular, ocular, gastrointestinal, vascular, and neurological involvements. The aim of present study is to assess pan immune inflammation value (PIN) value in BD in comparison to healthy control ,assess the PIN value in association with demographics and clinical characteristics of Behcet patients and to assess the PIN value in association with disease activity.

DETAILED DESCRIPTION:
Behçet's disease (BD) is a systemic vasculitis affecting both small and large blood vessels in the venous and arterial systems. It is a multiorgan disease with various manifestations, including mucocutaneous, articular, ocular, gastrointestinal, vascular, and neurological involvements. Inflammation of the vascular wall is the primary pathophysiology contributing to thrombosis in BD. Hematological and biochemical values are altered due to systemic inflammation and aberrant immune response. Neutrophils, lymphocytes, and platelets play a significant role in systemic inflammation and thrombosis. In addition to the number and volume of peripheral cells, changes in multiple cell count ratios, such as the platelet-to-lymphocyte ratio (PLR), neutrophil-to-lymphocyte ratio (NLR), and monocyte-to-lymphocyte ratio (MLR), have become important predictors of the diagnosis, disease activity, s and severe organ damage in rheumatologic disorders. pan immune inflammation value (PIV) was first described by Fuca et al and used to evaluate the inflammation. Literature showed that PIV performed better than previous immune-inflammatory biomarkers, such as NLR in colorectal cancer patients. PIV is calculated from four blood cell counts, including neutrophils, platelets, monocytes, and lymphocytes. In some rheumatological diseases such as RA, familial Mediterranean fever, and vasculitis, PIV has been studied.

In clinical practice, hematological and inflammatory laboratory tests are easily accessible and cost-effective. It is important to determine which blood parameter will be more effective in detecting disease activity and monitoring the treatment response in BD. In our study, our aim is to investigate the association of PIN with demographics and clinical characteristics of BD patients and its correlation with disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult BD patients who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease .
* Accept to participate in the current study.

Exclusion Criteria:

* Individuals with other autoimmune diseases.
* Patients unwilling to participate in the study.
* Patients less than 18 years old.
* Patients with malignancy or infections.
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult BD patients who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease attending Rheumatology, Rehabilitation and Physical Medicine Department, Assiut University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pan immune inflammation value (PIN value) in BD in comparison to healthy control | 3 months
  Using the ratio of neutrophil, monocyte, and platelet counts to lymphocyte count, NLR, MLR, and PLR were calculated. The pan immune inflammation value (PIV) was calculated by multiplying the neutrophil count (109/L) by the platelet count (109/L) and the monocyte count (109/L), and then dividing the result by the lymphocyte count (109/L).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Farrag, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yazici Y, Hatemi G, Bodaghi B, Cheon JH, Suzuki N, Ambrose N, Yazici H. Behcet syndrome. Nat Rev Dis Primers. 2021 Sep 16;7(1):67. doi: 10.1038/s41572-021-00301-1. PMID 34531393
- [Background] Bettiol A, Prisco D, Emmi G. Behcet: the syndrome. Rheumatology (Oxford). 2020 May 1;59(Suppl 3):iii101-iii107. doi: 10.1093/rheumatology/kez626. PMID 32348523
- [Background] Fuca G, Guarini V, Antoniotti C, Morano F, Moretto R, Corallo S, Marmorino F, Lonardi S, Rimassa L, Sartore-Bianchi A, Borelli B, Tampellini M, Bustreo S, Claravezza M, Boccaccino A, Murialdo R, Zaniboni A, Tomasello G, Loupakis F, Adamo V, Tonini G, Cortesi E, de Braud F, Cremolini C, Pietrantonio F. The Pan-Immune-Inflammation Value is a new prognostic biomarker in metastatic colorectal cancer: results from a pooled-analysis of the Valentino and TRIBE first-line trials. Br J Cancer. 2020 Aug;123(3):403-409. doi: 10.1038/s41416-020-0894-7. Epub 2020 May 19. PMID 32424148